CLINICAL TRIAL: NCT03139838
Title: Behavioral Economic Approaches to Improve Palliative Care for Critically Ill Patients
Brief Title: Prognosticating Outcomes and Nudging Decisions With Electronic Records in the ICU Trial
Acronym: PONDER-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Wake Forest University Health Sciences (Other); Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPenn IRB #826933; 52635 (Other Grant/Funding Number: Patrick and Catherine Weldon Donaghue Foundation)
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Critical Illness
Keywords: Palliative Care; Pragmatic Clinical Trial; Electronic Health Records; Economics, Behavioral
MeSH Terms: conditions — Critical Illness; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EHR-Based Intervention A (Active Comparator): Intervention A (Prognostication) will be an EHR-based screen prompt triggered for eligible patients. The intervention will consist of no more than two questions that can be completed in two minutes or less. Completion of the prompt will be encouraged but not required, and adherence will be assessed in a minimally intrusive manner.
  Interventions: Behavioral: EHR-Based Intervention A
- EHR-Based Intervention B (Active Comparator): Intervention B (Accountable Justification) will be an EHR-based screen prompt triggered for eligible patients. The intervention will consist of no more than two questions that can be completed in two minutes or less. Completion of the prompt will be encouraged but not required, and adherence will be assessed in a minimally intrusive manner.
  Interventions: Behavioral: EHR-Based Intervention B
- Combined EHR-Based Intervention (A+B) (Active Comparator): Intervention A and B prompts will be combined and triggered for eligible patients simultaneously. Completion of the prompt will be encouraged but not required, and adherence will be assessed in a minimally intrusive manner.
  Interventions: Behavioral: EHR-Based Intervention A; Behavioral: EHR-Based Intervention B
- Pre-Intervention (Control) (No Intervention): There is no trial-driven approach to care. All hospitals contribute a minimum of 5 months of outcomes data prior to adopting the intervention. Pre-specified outcomes data will be electronically extracted for patients meeting eligibility criteria but there will be no attempt to influence delivery of usual care within the hospital. The length of the control phase will differ at each hospital, dependent on the sequence in which hospitals are assigned to switch to the intervention phase.

INTERVENTIONS:
Behavioral: EHR-Based Intervention A — Intervention A will be a prompt for clinicians to document an estimated prognosis for patients at 6 months, and an assessment of predicted functional outcome if expected to survive.
  Other Names: Prognostication
  Arms: Combined EHR-Based Intervention (A+B); EHR-Based Intervention A
Behavioral: EHR-Based Intervention B — Intervention B will entail a prompt for clinicians to provide a reason for not offering patients and their families the alternative of care focused entirely on comfort despite recommendations from critical care professional societies to do so for patients at high risk for death or severely impaired functional recovery.
  Other Names: Accountable Justification
  Arms: Combined EHR-Based Intervention (A+B); EHR-Based Intervention B

SUMMARY:
This is a pragmatic, stepped-wedge, cluster randomized trial testing the real-world effectiveness of two different electronic health record (EHR) behavioral interventions in improving a number of patient- and family-centered processes and outcomes of care among seriously ill hospitalized patients. The investigators hypothesize that outcomes can be improved without raising costs by requiring intensive care unit clinicians to (i) document a prognostic estimate and (ii) provide a justification if they choose not to offer patients the option of comfort-oriented care. To test this hypothesis the investigators will conduct a 33-month trial at 17 intensive care units in 10 hospitals using the same Cerner EHR within Atrium Health System.

DETAILED DESCRIPTION:
The PONDER-ICU trial aims to generate large-scale, experimental evidence regarding the real-world effectiveness of two different electronic health record (EHR) behavioral interventions in improving a number of patient- and family-centered processes and outcomes of care among seriously ill hospitalized patients. The interventions are designed to increase intensive care unit (ICU) physicians' and advanced practitioners' (physician assistants and nurse practitioners) engagement of critically ill patients and caregivers in discussions about alternative treatment options, including care focused on comfort. To achieve this goal, the investigators will conduct a 33-month pragmatic, stepped-wedge cluster randomized clinical trial at 17 ICUs within 10 Atrium Health System hospitals. The investigators hypothesize that outcomes can be improved without raising costs by requiring ICU clinicians to (i) document a prognostic estimate (Intervention A) and (ii) provide a justification if they choose not to offer patients the option of comfort-oriented care (Intervention B). Approximately 4,750 adult patients (1) with chronic life-limiting illness and receiving continuous mechanical ventilation for ≥48 hours will be enrolled. Participating hospitals will be randomized into 5 clusters of 2 hospitals each. Each hospital will first contribute a minimum of 5 months of data collection during usual care in a control phase. Then, using the step-wedge design, all hospitals will implement the two EHR-based interventions. The order in which the interventions will be adopted and the timing of adoption at each hospital will both be determined by random assignment. After 12 months of utilizing Intervention A or Intervention B, each hospital will adopt and implement the second intervention in combination with the other. By the end of the trial, all hospitals will have utilized the combined interventions for at least 4 months. The primary outcome is a composite measure of hospital length of stay and mortality. Secondary outcomes include an array of clinical outcomes, as well as palliative care-related process measures.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old; AND
2. Admitted to 1 of the 17 participating ICUs; AND
3. Receipt of continuous mechanical ventilation for ≥ 48 hours (without interruption); AND
4. ≥ 1 life-limiting illness present on admission (ICD-9/10 code or discrete medical history data from EHR in prior 12 months):

   1. Chronic obstructive pulmonary disease
   2. Cirrhosis
   3. Congestive heart failure
   4. Dementia (all types)
   5. End-stage renal disease
   6. Hematologic malignancy
   7. Metastatic malignancy
   8. Motor neuron disease
   9. Pulmonary fibrosis
   10. Solid organ malignancy

Exclusion Criteria:

1) Patients younger than 18 years old are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Composite Measure: Length of Stay and In-Hospital Mortality | Duration of hospital stay, an expected average of 16 days
  The primary outcome is a composite measure of hospital length-of-stay and mortality that ranks deaths along the length-of-stay distribution

SECONDARY OUTCOMES:
Change in code status | Duration of hospital stay, an expected average of 16 days
  Change in documented code status during hospital admission
Initiation of additional forms of life-support | Duration of hospital stay, an expected average of 16 days
  Initiation of additional form of life-support (e.g. surgical feeding tube, dialysis) during hospital admission
Palliative care consult | Duration of hospital stay, an expected average of 16 days
  Receipt of palliative care consult during hospital admission
Time to palliative care consult | Duration of hospital stay, an expected average of 16 days
  The number of hours from ICU admission to inpatient palliative care consult
Palliative withdrawal of mechanical ventilation | Duration of hospital stay, an expected average of 16 days
  Palliative withdrawal of mechanical ventilation during hospital admission
Receipt of cardiopulmonary resuscitation (CPR) | Duration of hospital stay, an expected average of 16 days
  CPR prior to death or discharge
ICU mortality | Duration of hospital stay, an expected average of 16 days
  ICU mortality
ICU length of stay | Duration of hospital stay, an expected average of 16 days
  ICU length of stay (hours)
ICU readmission | Duration of hospital stay, an expected average of 16 days
  Readmission to an ICU within the same hospitalization
Duration of mechanical ventilation | Duration of hospital stay, an expected average of 16 days
  Hours of mechanical ventilation during hospital admission
Time to withdrawal of life-support | Duration of hospital stay, an expected average of 16 days
  The number of hours from trial enrollment to time that comfort-care order is placed
Hospital discharge disposition | Duration of hospital stay, an expected average of 16 days
  Hospital discharge disposition to home, hospice, long-term acute care, nursing facility, or rehabilitation
Quality of Dying & Death (1-item) | 48-72 hours following an in-hospital death
  Nurse-reported postmortem rating of a patient's dying experience
30-day hospital readmission | 30 days
  30-day hospital readmission
90-day hospital readmission | 30 days
  30-day hospital readmission
180-day hospital readmission | 30 days
  30-day hospital readmission
30-day mortality | 30 days
  Mortality rate at 30 days
90-day mortality | 90 days
  Mortality rate at 90 days
180-day mortality | 180 days
  Mortality rate at 180 days
Hospital free days | 180 days
  Hospital free days within 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, PhD, MD, Principal Investigator — University of Pennsylvania
Locations (10):
- United States (10):
  - Carolinas HealthCare System Stanly, Albemarle, North Carolina
  - Carolinas HealthCare System, NorthEast, Charlotte, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Atrium Health CMC-Mercy, Charlotte, North Carolina
  - Atrium Health Pineville, Charlotte, North Carolina
  - Atrium Health University City, Charlotte, North Carolina
  - Atrium Health Lincoln, Lincolnton, North Carolina
  - Atrium Health Union, Monroe, North Carolina
  - Carolinas HealthCare System Blue Ridge-Morganton, Morganton, North Carolina
  - Atrium Health Cleveland, Shelby, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courtright KR, Singh J, Dress EM, Bayes B, Harhay MO, Chowdhury M, Lu Y, Lee KM, Small DS, Whitman C, Tian J, Madden V, Hetherington T, Placket L, Sullivan DM, Burke HL, Green MB, Halpern SD. Nudging Clinicians to Promote Serious Illness Communication for Critically Ill Patients: A Pragmatic Cluster Randomized Trial. JAMA Intern Med. 2025 May 1;185(5):510-520. doi: 10.1001/jamainternmed.2025.0090. PMID 40094649
- [Derived] Courtright KR, Dress EM, Singh J, Bayes BA, Chowdhury M, Small DS, Hetherington T, Plickert L, Detsky ME, Doctor JN, Harhay MO, Burke HL, Green MB, Huynh T, Sullivan DM, Halpern SD; PONDER-ICU Investigative Team. Prognosticating Outcomes and Nudging Decisions with Electronic Records in the Intensive Care Unit Trial Protocol. Ann Am Thorac Soc. 2021 Feb;18(2):336-346. doi: 10.1513/AnnalsATS.202002-088SD. PMID 32936675